CLINICAL TRIAL: NCT04942028
Title: Randomized Controlled Trial of Internet-delivered Exposure-based Treatment vs. Standardized Education for Distress Related to Somatic Symptoms in Primary Care
Brief Title: Exposure Therapy vs. Standardized Education for Distress Related to Somatic Symptoms
Acronym: SOMEX1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-01400
Record Dates: First submitted 2021-06-17; First posted 2021-06-28 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Somatic Symptom and Related Disorders; Medically Unexplained Symptoms; Psychological Factors Affecting Other Medical Conditions
Keywords: exposure; primary care
MeSH Terms: conditions — Medically Unexplained Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered exposure-based treatment (Experimental): 10 weeks of therapist-guided exposure-based treatment delivered via the Internet.
  Interventions: Behavioral: Exposure
- Internet-delivered standardized education and prolonged assessment (Active Comparator): 10 weeks of therapist-guided intervention based on prolonged assessment and routine care educational material delivered via the Internet.
  Interventions: Behavioral: Standardized education; Behavioral: Prolonged assessment

INTERVENTIONS:
Behavioral: Exposure — Systematic confrontation with stimuli associated with symptom-related distress, to achieve therapeutic changes in cognitions or behavior
  Arms: Internet-delivered exposure-based treatment
Behavioral: Standardized education — Standardized routine care education for individuals suffering from distress related to somatic symptoms, primarily focusing on healthy lifestyle behaviors such as sleep, diet, and exercise
  Arms: Internet-delivered standardized education and prolonged assessment
Behavioral: Prolonged assessment — Patients are encouraged to keep a rudimentary symptom diary to track if and how their symptoms interact with mood and lifestyle behaviors
  Arms: Internet-delivered standardized education and prolonged assessment

SUMMARY:
The annual societal cost of medically unexplained symptoms in Sweden is approximately 40 billion SEK, i.e., similar to the annual cost of cancer. Prevalent chronic diseases like asthma and diabetes are also commonly associated with somatic symptoms that lead to significant distress and pervasive behavioral changes that result in functional impairment and place added strain on the health care system. Exposure-based treatment, where the patient willingly engages with stimuli that give rise to unwanted physical sensations or distress, has shown promise in reducing somatic symptom load and increasing quality of life in several conditions where patients commonly report substantial distress related to somatic symptoms, such as in asthma, musculoskeletal pain, and functional gastrointestinal syndromes. In routine care, however, access to such exposure-based treatment is limited. One reason for this is probably that there exists no flexible exposure-based treatment protocol that can be easily tailored to suit a wide spectrum of patient groups who suffer from distress related to recurrent somatic symptoms. In a recent single group feasibility trial (N=33) at Karolinska Institutet, Sweden, the investigators found that such a tailored exposure-based treatment delivered in an online text-based format can be acceptable, with high treatment adherence, adequate treatment satisfaction, large and lasting within-group improvement, and no serious adverse events. This is a randomized controlled trial (N=160) where the investigators aim to test if the same tailored internet-delivered exposure-based treatment is more efficacious than a standardized education control for adult patients with clinically significant distress related to somatic symptoms in a primary care setting. Primary outcome is change in self-rated somatic symptom burden as modelled using linear mixed models fitted on weekly Patient Health Questionnaire 15 sum scores over the treatment period. Long-term efficacy is assessed up to one year after treatment and cost-effectiveness is investigated based on the incremental cost-effectiveness ratio.

DETAILED DESCRIPTION:
Approximately one fifth of primary care patients seek care for symptoms that cannot readily be given a medical explanation. In addition, primary care is tasked with offering care for prevalent chronic diseases such as asthma and diabetes where somatic symptoms often lead to distress and pervasive behavioral changes. Though a concern with somatic symptoms can be fully warranted, helpful, and transient, it can also be persistent and lead to much unnecessary suffering. Existing treatments commonly yield insufficient effects on medically unexplained symptoms.

Psychological factors - in particular the preoccupation with symptoms - have been found to affect the perception and intensity of a large number of physical symptoms, both with and without a clear medical genesis. In pain, it has for example been found that fear and the preoccupation with symptoms can have a more substantial predictive value for chronicity than pain itself. In general, in individuals who suffer from clinically significant symptom preoccupation, behaviors intended to evaluate symptoms, seek information about symptoms, or avoid discomfort have been found to often contribute to worsened function and increased symptom burden in the long term.

This makes exposure, where the patient willingly and systematically approaches stimuli that give rise to unwanted symptoms or discomfort while refraining from acting on symptoms, a logical intervention. There are several examples where exposure-based treatment has been found to be efficacious when protocols were written to suit a particular group of patients where distress associated with somatic symptoms is common, e.g., a particular functional somatic syndrome in terms of fibromyalgia and irritable bowel syndrome, or a chronic somatic condition such as asthma or atrial fibrillation. Typically, effects on symptoms and the preoccupation with symptoms have been large, and there is evidence to suggests that a reduction in somatic symptom burden may have been mediated by a reduction in symptom preoccupation or behaviors that serve to reduce distress in the short term.

Generalist primary care clinics typically do not have the resources necessary for administering specific psychological treatments for a large number specific functional somatic syndromes or chronic somatic conditions. The investigators suspect that a more general treatment protocol that can be tailored to suit a wide spectrum of physical symptoms could dramatically improve access to exposure-based treatment for patients with distress related to somatic symptoms. This may be particularly true if treatment can be delivered via the internet, which requires less therapist time but often results in similar effects as face-to-face treatment.

The investigators recently completed a feasibility trial at Karolinska Institutet, Sweden (NCT04511286), where the investigators found that an internet-delivered flexible exposure-based treatment for individuals with high levels of symptom preoccupation regardless of somatic symptom domain (N=33; e.g., functional gastrointestinal symptoms, atrial fibrillation, migraine) can be delivered with high treatment adherence, adequate client satisfaction, large and lasting improvement in self-reported somatic symptoms and symptom preoccupation, and no serious adverse events. It is thus motivated to evaluate this treatment format further.

In further evaluating the flexible exposure-based treatment approach for patients with distress related to somatic symptoms it is imperative to conduct a randomized controlled trial versus an informative control condition, focusing on effects on somatic symptoms and symptom preoccupation. It is also important to evaluate if the treatment can be effective in a routine clinical setting and when patients are referred via a clinician such as a general practitioner. In this trial, the investigators aim to evaluate if flexible internet-delivered exposure-based treatment is more effective than an internet-delivered standardized routine care education program for patients with distress related to somatic symptoms in primary care.

* Primary research question:

Compared to the control condition, does flexible internet-delivered exposure-based treatment lead to a larger average improvement in self-rated somatic symptom burden as assessed using the Patient Health Questionnaire 15 (PHQ-15)? Hypothesis: Yes.

* Key secondary research questions:

Compared to the control condition, does flexible internet-delivered exposure-based treatment lead to a larger average improvement in symptom preoccupation, psychiatric symptom burden, and functional impairment? Hypothesis: Yes.

In flexible internet-delivered exposure-based treatment, are effects typically maintained up to 12 months after treatment? Hypothesis: Yes.

Is flexible internet-delivered exposure-based treatment cost-effective compared to the control condition? Hypothesis: Yes.

Is the controlled effect of the flexible exposure-based treatment on self-rated somatic symptoms moderated by baseline symptoms and preoccupation? Hypothesis: Yes.

Is the effect of the flexible exposure-based treatment on self-rated somatic symptom burden mediated by a reduction in symptom preoccupation? Hypothesis: Yes.

ELIGIBILITY:
Inclusion Criteria:

* (i) Either much bothered by at least one somatic symptom (2 points on at least one item of the PHQ-15) or at least a moderate overall somatic symptom burden (PHQ-15 sum ≥10), with (ii) recurrent distress related to somatic symptoms ≥4 months
* Interested in completing an intense psychological treatment with the aim of reducing distress associated with physical symptoms
* Adult (≥18 years old)
* Living in Stockholm County
* Can read and write in Swedish
* Complete baseline assessment

Exclusion Criteria:

* Symptoms best explained by, or clinical picture dominated by, severe health anxiety or a non-somatoform psychiatric disorder such as depression, panic disorder, primary insomnia, a chronic stress disorder, or an acute stress disorder
* Severe psychiatric condition or suicidal ideation
* Clear medical risk in taking part in exposure-based treatment (e.g., pregnancy) or somatic condition (e.g., recent cancer diagnosis), or treatment for somatic condition (e.g., recent chemotherapy), makes treatment unfeasible
* Continuous psychotropic medication (antidepressants, anticonvulsants, mood-stabilizers, antipsychotics) not stable in past 4 weeks, or not expected to remain stable over the main phase of the trial
* Severe alcohol or substance use disorder likely to interfere with treatment
* Planned absence for more than 1 week during the intended main phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-15 (PHQ-15) | Change over the main phase, as modelled using data from all 11 assessments from the baseline assessment to the primary endpoint (≤45 days after treatment). Secondary analyses incorporate 6- and 12-months follow-up assessments.
  Theoretical range: 0-30. A higher score indicates a higher subjective somatic symptom burden.

SECONDARY OUTCOMES:
Somatic Symptom Disorder-B Criteria Scale (SSD-12) | Change over the main phase, as modelled using data from all 11 assessments from the baseline assessment to the primary endpoint (≤45 days after treatment). Additional analyses incorporate 6- and 12-months follow-up assessments.
  Theoretical range: 0-48. A higher score indicates higher degree of preoccupation with symptoms.
Symptom Preoccupation Scale (preliminary scale) | Change over the main phase, as modelled using data from all 11 assessments from the baseline assessment to the primary endpoint (≤45 days after treatment). Additional analyses incorporate 6- and 12-months follow-up assessments.
  Under development. A higher score indicates higher degree of preoccupation with symptoms.
GAD-7 | Change over the main phase, as modelled using data from the baseline assessment and primary endpoint (≤45 days after treatment). Additional analyses incorporate 6- and 12-months follow-up assessments.
  Theoretical range: 0-21. A higher score indicates more general anxiety.
Patient Health Questionnaire (PHQ-9) | Change over the main phase, as modelled using data from the baseline assessment and primary endpoint (≤45 days after treatment). Additional analyses incorporate 6- and 12-months follow-up assessments.
  Theoretical range: 0-27. A higher score indicates more symptoms of depression.
12-item WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | Change over the main phase, as modelled using data from the baseline assessment and primary endpoint (≤45 days after treatment). Additional analyses incorporate 6- and 12-months follow-up assessments.
  Theoretical range: 0-100. A higher score indicates more disability.
14-item Health Anxiety Inventory (HAI-14) | Screening only
  Theoretical range: 0-42. A higher score indicates more health anxiety.
Alcohol Use Disorders Identification Test (AUDIT) | Screening only
  Theoretical range: 0-40. A higher score indicates more problematic alcohol use.
Drug Use Disorders Identification Test (DUDIT) | Screening only
  Theoretical range: 0-44. A higher score indicates more problematic substance use.
Credibility/Expectancy scale (C/E scale) | Week 3 of main phase
  Theoretical range: 0-50. A higher score indicates higher credibility/expectancy.
Working Alliance Inventory (WAI) | Week 3 of main phase
  Theoretical range: 6-42. A higher score indicates better relationship with the therapist.
Client Satisfaction Questionnaire (CSQ-8) | Primary endpoint assessment (≤45 days after treatment)
  Theoretical range: 8-32. A higher score indicates higher satisfaction with treatment.
EuroQol 5D (EQ-5D) | Data from the baseline assessment, the primary endpoint, and the 6- and 12-month follow-up are used for health economic analysis focusing on the main phase.
  Theoretical range: 0-1, i.e., scored as utility for the purpose of calculating quality-adjusted life years for health economic analysis. A higher utility score indicates a higher health-related quality of life.
Trimbos Institute and Institute of Medical Technology Questionnaire for Costs Associated with Psychiatric Illness (TIC-P) | Data from the baseline assessment, the primary endpoint, and the 6- and 12-month follow-up are used for health economic analysis focusing on the main phase.
  This instrument is scored in terms of resource use for the purpose of calculating societal costs for health economic analysis.
Four questions corresponding to presumed components of subjective somatic symptom burden | Measured at screening, baseline assessment, and the primary endpoint
  These questions concern (1) somatic symptom severity, (2) somatic symptom frequency/duration, (3) distress related to somatic symptoms, and (4) the impact of somatic symptoms on disability. Answers are given on visual analogue scales.
Seven questions probing into basic emotions related to somatic symptoms | Measured at screening, baseline assessment, and the primary endpoint
  Answers are given on visual analogue scales.

CONTACTS AND LOCATIONS:
Overall Officials: Erland Axelsson, PhD, Principal Investigator — Liljeholmen academic primary care clinic, Region Stockholm
Locations (1):
- Liljeholmen academic primary care clinic, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
We are willing to consider reasonable requests for individual participant data (IPD) and to consult the responsible parties. However, we do not expect to be granted permission to share IPD as long as, under Swedish and European Union (EU) data protection and privacy legislation, the IPD constitutes personal data meaning that it is possible to, using the existing study database, link the IPD to an identifiable living natural person. Ten years after the last publication, the information necessary for individuals to be identified will be deleted and documentation from the trial will be archived for long-term storage. We expect to include anonymized IPD in this archive. It is our understanding that, under EU law, IPD without the existence of information necessary for individuals to be identified does not constitute personal because the IPD can no longer be linked to a living natural person. Thus, 10 years after the last publication and onwards, we expect to be able to share IPD on request.

REFERENCES:
- See also: Simple exposure protocol administered over 10 weeks — https://osf.io/b8hev/

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Study protocol with rudimentary SAP (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT04942028/Prot_SAP_001.pdf
  • Statistical Analysis Plan: Detailed SAP for primary publication (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT04942028/SAP_002.pdf
  • Statistical Analysis Plan: Detailed SAP for secondary analysis of cost-effectiveness (2025-03-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT04942028/SAP_003.pdf
  • Statistical Analysis Plan: Detailed SAP for secondary analysis of mediators (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT04942028/SAP_004.pdf